CLINICAL TRIAL: NCT06176846
Title: Effect of Immersive Virtual Reality Exergaming Program on Physical Fitness, Functional Capacity and Physical Activity In Adolescents Diagnosed With Juvenile Idiopathic Arthritis: A Randomized Controlled Study
Brief Title: Immersive Virtual Reality Exergaming Program in Adolescents Diagnosed With Juvenile Idiopathic Arthritis
Acronym: JiaFiT-XR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assoc.Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1795570
Record Dates: First submitted 2023-12-01; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Exercise; Exergaming; Physical Fitness
MeSH Terms: conditions — Arthritis, Juvenile; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality Exergaming Group (Experimental): Patients in this group will be included in an exergaming program using Oculus Quest 3 glasses.
  Interventions: Behavioral: Immersive Virtual Reality Exergaming Program
- Home-Based Exercise Group (Experimental): Patients in this group will be included in a home-based exercise program.
  Interventions: Behavioral: Home-Based Exercise Program

INTERVENTIONS:
Behavioral: Immersive Virtual Reality Exergaming Program — Oculus Quest 3 glasses will be used as hardware for the IVR exergame program, and "Boxing", "HIIT", "Combat", "Sculpt" and Dance, among the Fit-XR games that offer virtual reality experience for fitness, will be selected according to the physical fitness level of the subjects and personalized multicomponent ( balance, strength, agility, endurance) IVR exergame program will be created. The exercise program is limited to 25-30 minutes a day and will be applied 2 days a week for 8 weeks in the clinic under the supervision of a physiotherapist. The exergaming program will be progressed according to the difficulty level, duration and technical characteristics of the games.
  Arms: Immersive Virtual Reality Exergaming Group
Behavioral: Home-Based Exercise Program — In the home-based exercise program, a personalized multicomponent (balance, strength, agility, endurance) exercise program will be applied according to the physical fitness level of the subjects. The exercises will progress by increasing the difficulty level and number of repetitions of the exercises. An e-brochure will be given to the subjects for the exercises, the exercises will be shown to the subjects on the 1st day, and exercise control will be carried out in the 1st week and the 4th week.
  Arms: Home-Based Exercise Group

SUMMARY:
The aim of the study is to investigate the effect of home-based exercise program versus personalized IVR exergame (Fit-XR) program on physical fitness, functional capacity and physical activity in adolescents with Juvenile idiopathic arthritis. Patients followed up by four tertiary pediatric rheumatology centers will be included in the project. Two different exercise programs will be applied to the patients by experienced physiotherapists. Fit-XR program will be 25-30 minutes a day and will be applied 2 days a week for 8 weeks under the supervision of a physiotherapist in the clinic. The total points obtained by the participants during the FiT-XR games will be recorded after each training session. In the second group, a personalized multicomponent (balance, strength, agility, endurance) home- based exercise program will be applied according to the physical fitness level of the children.

ELIGIBILITY:
Inclusion Criteria:

* Having a definitive diagnosis of JIA according to the ILAR classification at least 6 months ago
* Being between the ages of 13-18

Exclusion Criteria:

* JIA diagnosis was made less than a month ago
* Having had a surgical or arthroscopic operation within the last year
* Presence of active synovitis or arthritis
* Have a disease that may limit the ability to exercise or increase the cardiovascular risk of exercise, including cardiovascular, pulmonary, musculoskeletal, or metabolic disorders
* Having active vestibular disease
* Having a neurological disease that prevents walking and exercising
* Having been exercising regularly for the last 6 months
* Having severe vision and hearing problems
* Use of any medication or supplement known to increase anabolic responses
* Having mental inability to understand the exercises

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
FitnessGram Physical Activity Test Battery-Progressive Aerobic Cardiovascular Endurance Running (PACER) | Change from Baseline FitnessGram Physical Activity Test Battery-Progressive Aerobic Cardiovascular Endurance Running (PACER) at 8 weeks
  PACER is an adapted version of the 20 meter shuttle run test and is a field test consisting of multiple stages. The participant will run back and forth in a 20 meter area accompanied by the music coming from the voice recorder. The beep indicates when the participant should finish a lap. The test will start at slow speeds and will gradually increase each minute. The test will be terminated when the participant cannot continue to run at the level he has reached. The number of laps completed at the end of the test will be recorded. PACER is a more fun alternative to other distance running tests. It is recommended for use in children, adolescents and young adults. PACER will be used to assess the aerobic capacity of adolescents.
6 Minute Walk Test (6 MWT) | Change from Baseline 6 Minute Walk Test (6 MWT) at 8 weeks
  The 6-minute walk test is a well-tolerated, easy-to-apply and simple test that shows the submaximal level of functional capacity. This test measures the distance that participants can walk quickly on a hard and flat surface in 6 minutes. Participants rest in a chair near the starting position for at least 10 minutes before the start of the test. Before and after the test, heart rate, blood pressure, saturation are measured, and fatigue level is determined with the Modified Borg scale. Participants are told how to perform the test. At the end of the test, the distance walked by the participants in 6 minutes will be recorded in meters. The 6 Minute Walk Test will be used to evaluate the functional capacities of adolescents.
30 second sit to stand test (30SST) | Change from Baseline 30 second sit to stand test (30SST) at 8 weeks
  30 second sit to stand test is commonly used for assessing lower limb's functional capacity. Participants are asked to rise from a seated position and sit as quickly and safely as possible in 30 s. The completed number of chair stands within 30 s is counted and recorded for this test. Arms are crossed at the wrists and held against the chest. Feet place on the floor at an angle slightly back from the knees. The participant starts with "go" word and rose to a full stand and then returned to the initial seated position. The participants are encouraged to complete as many full stands as possible within a 30-second time limit. 30 second sit to stand test will be used to evaluate tower limb's functional capacity of the adolescents.

SECONDARY OUTCOMES:
FitnessGram Physical Activity Test Battery-Bioelectrical Impedance Analysis | Change from Baseline FitnessGram Physical Activity Test Battery-Bioelectrical Impedance Analysis at 8 weeks
  BIA is based on the principle of measuring resistance to the flow of a low-level electric current through the body. In our study, body composition parameters such as muscle, fat and water ratio will be evaluated with the Tanita SC240 device.
FitnessGram Physical Activity Test Battery-Curl-up Test | Change from Baseline FitnessGram Physical Activity Test Battery-Curl-up Test at 8 weeks]
  The participant will begin the test in the supine position, knees flexed approximately 140 degrees, feet flat on the floor, and legs slightly apart. The participant's arms will be parallel to the floor and torso. The palm will be positioned on the floor with the fingers stretched out. The purpose of this test is to do as many sit-ups as possible at a given speed. A maximum of 75 shuttles counts. The number of shuttles performed at the end of the test will be recorded. The curl-up test will be used to evaluate the abdominal muscle strength and endurance of adolescents.
FitnessGram Physical Activity Test Battery-Trunk Lift Test | Change from Baseline FitnessGram Physical Activity Test Battery-Trunk Lift Test at 8 weeks
  The participant will begin the test in the prone position with their hands placed under the thigh. A sign will be placed on the floor at the participant's eye level. During the movement, the participant will focus on this sign. During the test, the participant slowly and in a controlled manner raises their torso to a maximum height of 12 inches. The head is kept in neutral alignment with the spine. At the end of the test, the distance between the floor and the participant's chin will be measured with a ruler and the score will be recorded in centimeters (cm). Trunk lift test will be used to evaluate trunk extensor muscle strength and flexibility of adolescents
FitnessGram Physical Activity Test Battery-Push-up Test | Change from Baseline FitnessGram Physical Activity Test Battery-Push-up Test at 8 weeks
  The participant will begin the test in the prone position, with their hands shoulder-width or wider than shoulder-width apart, fingers stretched, palms on the floor, and legs slightly apart. During the test, the participant lowers his torso towards the ground and raises himself up again when his elbows are bent 90º. The movement is repeated as much as possible. The rhythm is set to 20 push-ups per minute or 1 push-up per 3 seconds. The test is terminated when the participant makes a mistake twice. The number of push-ups performed at the end of the test will be recorded. The push-up test will be used to evaluate the upper extremity muscle strength and endurance of adolescents.
Physical Activity Test Battery-Back Saver Sit and Reach Test | Change from Baseline FitnessGram Physical Activity Test Battery-Back Saver Sit and Reach Test at 8 weeks
  During the test, the participant takes off his shoes and sits in front of the test apparatus. A box is needed for the test. This box is 35 cm long, 45 cm wide, 32 cm high. A top plate 55 cm long and 45 cm wide is put on top of the box. One leg of the participant is completely straight while the other is bent at the knee. The participant reaches forward four times with their hands on top of each other, holding the fourth reach position for 1 second. At the end of the test, the distance traveled will be recorded. The Back Saver Sit and Reach Test will be used to evaluate the hamstring flexibility of adolescents.
Physical Activity-Heart rate for daily living activities | Change from Baseline heart rate during daily living activities at 8 weeks
  The adolescents included in the study will be given a smart watch and will be asked to use the watches for 8 weeks. The data obtained on physical activity behaviors of adolescents for 2 months through smart watches will be transferred to the cloud and web platform with the mobile application. With wearable activity tracker watches, data on the person's heart rates during the daily living activities will be recorded and transferred to the cloud.
Physical Activity-The number of steps taken per day | Change from the number of steps taken per day at 8 weeks
  The adolescents included in the study will be given a smart watch and will be asked to use the watches for 8 weeks. The data obtained on physical activity behaviors of adolescents for 2 months through smart watches will be transferred to the cloud and web platform with the mobile application. With wearable activity tracker watches, data on the person's number of steps taken per day will be recorded and transferred to the cloud.
Physical Activity-daily calories burned | Change from the daily calories burned at 8 weeks
  The adolescents included in the study will be given a smart watch and will be asked to use the watches for 8 weeks. The data obtained on physical activity behaviors of adolescents for 2 months through smart watches will be transferred to the cloud and web platform with the mobile application. With wearable activity tracker watches, data on the person's daily calories burned will be recorded and transferred to the cloud.
Physical Activity-daily oxygen consumption | Change from the daily oxygen consumption at 8 weeks
  The adolescents included in the study will be given a smart watch and will be asked to use the watches for 8 weeks. The data obtained on physical activity behaviors of adolescents for 2 months through smart watches will be transferred to the cloud and web platform with the mobile application. With wearable activity tracker watches, data on the person's daily oxygen consumption will be recorded and transferred to the cloud.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Assoc.Prof., Principal Investigator — Istanbul University-Cerrahpaşa, Faculty of Health Science, Department of Physiotherapy and Rehabilitation; Nuray Aktay Ayaz, Prof.Dr., Study Director — Istanbul Faculty of Medicine, Department of Internal Medicine, Department of Pediatric Rheumatology; Figen Cakmak, MD, Study Chair — Health Science University, Cam and Sakura City Hospital; Betul Sozeri, Prof.Dr., Study Chair — Health Science University, Umraniye Research and Training Hospital; Asena Yekdaneh, MSc, Pt, Study Chair — Istanbul University-Cerrahpasa, Institute of Postgraduate Education; Asya Albayrak, MSc, Pt, Study Chair — Istanbul University-Cerrahpasa, Institute of Postgraduate Education; Irem Donmez, PT, Study Chair — Istanbul University-Cerrahpasa, Institute of Postgraduate Education; Yusuf Acikgoz, PT, Study Chair — Istanbul University-Cerrahpaşa, Faculty of Health Science, Department of Physiotherapy and Rehabilitation
Locations (4):
- Turkey (Türkiye) (4):
  - Istanbul University Medical Faculty Hospital, Istanbul
  - Cam and Sakura City Hospital, Istanbul
  - Istanbul University-Cerrahpasa, Faculty of Health Science, Department of Physiotherapy and Rehabilitation, Istanbul
  - Umraniye Research and Training Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No